CLINICAL TRIAL: NCT07236346
Title: Effects of Parent-child Co-participation in Physical Activity on Physical Activity Levels and Motor Skills of Children With Autism Spectrum Disorder: a Quasi-experimental Study
Brief Title: Effects of Parent-child Co-participation in Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayburt University (Other)
Responsible Party: Principal Investigator, Erkan Yarımkaya, Assoc. Prof. Dr, Bayburt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: BU-SPBF-EY-01
Record Dates: First submitted 2025-11-13; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Autism Spectrum Disorder (ASD
Keywords: physical activity; parent; autism spectrum disorder; motor skills
MeSH Terms: conditions — Autism Spectrum Disorder; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The current study was a quasi-experimental study designed to determine the effectiveness of an 8-week PA intervention using two modes of delivery to improve PA levels and FMS in children with ASD. The quasi-experimental design is a frequently preferred research design, particularly in education research, where it is not possible to control all variables. A pre-test in the design helps determine the similarity of the groups before the intervention, while a post-test allows interpretation of the effects of the intervention on the participants.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- parent-child group (Experimental): This group included parental involvement. Parents and children engaged in PA together three days a week, each session lasting approximately one hour.
  Interventions: Behavioral: A parent-child co-participation in physical activity
- child group (Experimental): This group did not include parental involvement. Only children with ASD engaged in PA three days a week, each session lasting approximately 1 hour.
  Interventions: Behavioral: A parent-child co-participation in physical activity
- control group (No Intervention): This group continued their normal routines and activities throughout the intervention.

INTERVENTIONS:
Behavioral: A parent-child co-participation in physical activity — Parents in PCG-A engaged in PA with their children three days a week. All parents attended the sessions and engaged in partner warm-ups, partner functional exercises, partner games, and partner cool-downs with their children. Children in CG-B engaged in PA with their peers three days a week without parental involvement, engaging in partner warm-ups, partner functional exercises, partner games, and partner cool-downs. Both intervention groups were compared with a control group. We instructed the control group to maintain their normal routines and activities throughout the intervention and asked them to participate in a pre-test and post-test. A demonstration strategy was used to teach the activities. We provided immediate feedback to encourage and support children with ASD and their parents. We also chatted with the children and parents at the end of each daily physical activity session to evaluate the effectiveness of the session and prepare them for the next session.
  Arms: child group; parent-child group

SUMMARY:
Literature reviews and studies of physical activity (PA) interventions suggest that active parental involvement is an important component of supporting PA levels in children with autism spectrum disorders (ASD). Parents have also viewed these interventions as a valuable source of social support and motivation for themselves and their children with ASD; however, parents have reported a lack of PA interventions specifically involving parental involvement to increase PA levels in their children.

To our knowledge, only a handful of PA studies in the literature have examined PA levels or fundamentals movement skills (FMS) in children with ASD and have included parental involvement. Overall, findings from previous studies have shown that PA interventions that include parental involvement successfully improve PA levels and FMS in children with ASD. Given the potential benefits and the increasing interest in family-based interventions, supporting parent-child co-participation in PA may be a possible strategy to promote PA among children and parents. To date, studies on parent-child co-participation in PA have mostly focused on improving PA levels and FMS in children with ASD using web-based interventions such as social media, websites, and online systems. Furthermore, with the exception of two studies, the focus of these studies was on PA levels and not FMS in children with ASD. Furthermore, not all previous studies have created PA groups with and without parental involvement to explore whether parent-child co-participation truly makes a difference. We addressed these limitations in the current study and used a design that included a parent-child PA group, a child PA group, and a control group to examine both PA levels and FMS in children with ASD. Therefore, the purpose of this study was to examine the effects of parent-child co-participation on PA levels and FMS in children with ASD.

ELIGIBILITY:
Inclusion Criteria:

* willingness to participate in the study,
* being the primary guardian of a child with ASD between,
* having an ASD diagnosis confirmed GARS-2-TV,
* being between the ages of four and eleven,
* being able to walk independently.

Exclusion Criteria:

* those who do not attend at least one of the sessions of the training program,
* children with physical health problems (based on self-report and clinical diagnosis) will be excluded from the study.

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
The Leisure Time Exercise Questionnaire (LTEQ) | 8 weeks
  The Leisure Time Exercise Questionnaire (LTEQ) was used to assess children's PA levels before and after the intervention. The LTEQ consists of three questions that seek information on the number of times children engage in mild, moderate, and strenuous intensity PA for at least 15 minutes in a typical week.
  It was applied to the participants in the intervention groups twice, before and after 8 weeks.

SECONDARY OUTCOMES:
The Test of Gross Motor Development-3 (TGMD-3) | 8 weeks
  The TGMD-3 examines 13 gross motor skills, divided into two subsections: locomotor skills and ball skills. The TGMD-3 has been used in children with ASD aged 4 to 11 years. The TGMD-3 has been reported to have acceptable validity and reliability when measuring motor skills in ASD children. The TGMD-3 contains 3 to 5 criteria for each gross motor skill, which are integral to each other.
  It was applied to the participants in the intervention groups twice, before and after 8 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Work, Bayburt, Bayburt, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Since the study has not been published yet, I will fill in this section again when it is published.

REFERENCES:
- [Background] 1. American Psychiatric Association. Diagnostic and statistical manual of mental disorders. 5th ed. Washington DC: American Psychiatric Association; 2013.
- See also: Personal web site — https://bayburt.edu.tr/en/personel/erkan-yarimkaya-p1151